CLINICAL TRIAL: NCT06234722
Title: Modeling Tobacco Regulatory Impacts in Appalachia Using the Experimental Tobacco Marketplace
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mikhail N Koffarnus (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Mikhail N Koffarnus, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 87440; 1U54DA058256-01 (NIH)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use; Cigarette Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Mixed crossover-factorial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rural - Conventional Cigarette (Placebo Comparator): Participants who reside in rural locales of Appalachian KY and receive conventional cigarettes during the sampling period.
  Interventions: Behavioral: Reduced nicotine regulatory environment; Behavioral: Restriction on characterizing flavors in combustible nicotine products; Behavioral: Restriction on characterizing flavors in noncombustible nicotine products
- Peri-Urban - Conventional Cigarette (Placebo Comparator): Participants who reside in peri-urban locales of Appalachian KY and receive conventional cigarettes during the sampling period.
  Interventions: Behavioral: Reduced nicotine regulatory environment; Behavioral: Restriction on characterizing flavors in combustible nicotine products; Behavioral: Restriction on characterizing flavors in noncombustible nicotine products
- Peri-Urban - Very Low Nicotine Cigarette (Active Comparator): Participants who reside in peri-urban locales of Appalachian KY and receive very low nicotine cigarettes during the sampling period.
  Interventions: Drug: Very Low Nicotine Cigarette; Behavioral: Reduced nicotine regulatory environment; Behavioral: Restriction on characterizing flavors in combustible nicotine products; Behavioral: Restriction on characterizing flavors in noncombustible nicotine products
- Rural - Very Low Nicotine Cigarette (Active Comparator): Participants who reside in rural locales of Appalachian KY and receive very low nicotine cigarettes during the sampling period.
  Interventions: Drug: Very Low Nicotine Cigarette; Behavioral: Reduced nicotine regulatory environment; Behavioral: Restriction on characterizing flavors in combustible nicotine products; Behavioral: Restriction on characterizing flavors in noncombustible nicotine products

INTERVENTIONS:
Drug: Very Low Nicotine Cigarette — Participants will be assigned to one of two investigational cigarette nicotine levels for the duration of the experiment: 0.4mg/g or 15.8mg/g
  Arms: Peri-Urban - Very Low Nicotine Cigarette; Rural - Very Low Nicotine Cigarette
Behavioral: Reduced nicotine regulatory environment — In this regulatory environment, participants' usual combustible cigarette will not be available in the Experimental Tobacco Marketplace and only the participants' assigned investigational cigarette will be the only available combustible cigarette.
Behavioral: Restriction on characterizing flavors in combustible nicotine products — In this regulatory environment, menthol and other characterizing flavors in combustible nicotine products will not be available in the Experimental Tobacco Marketplace. Only tobacco or no flavored combustible nicotine products will be the only combustible nicotine products available.
Behavioral: Restriction on characterizing flavors in noncombustible nicotine products — In this regulatory environment, menthol and other characterizing flavors in noncombustible nicotine products will not be available in the Experimental Tobacco Marketplace. Only tobacco or no flavored noncombustible nicotine products will be the only noncombustible nicotine products available.

SUMMARY:
The goal of this project is to look at the effect of proposed tobacco product regulations in Appalachian Kentucky. Appalachian Kentucky is a diverse and underserved rural area that would benefit from more tobacco regulation research. Researchers will study the effects of three proposed tobacco product regulations among users of tobacco products in Appalachian KY. Researchers will also study how degree of rurality effects how those regulations impact behavior. Participants will be asked to complete online surveys and tests, online shopping sessions in a simulated Experimental Tobacco Marketplace, and track their tobacco product use throughout the 9-week experiment.

DETAILED DESCRIPTION:
After granting informed consent, participants will complete a baseline assessment session. This will be followed by an extended 9-week sampling period to acclimate participants to their randomly assigned experimental cigarette and allow any shifts in product consumption patterns to materialize. In the final week of this sampling period, participants will complete behavioral assessments and a series of assessments to assess the impact of potential regulatory environments relevant to our aims.

Experimental Tobacco Marketplace. In this procedure, participants will complete purchasing scenarios in our realistic tobacco/nicotine product marketplace to model and examine the impact of each of the proposed tobacco product regulations. Participants will be seated in front of a computer to access an online marketplace with an interface similar to many online merchants. This will allow participants to browse through the selection of products and add as many as they desire of each product to the virtual shopping cart. Each product will have the price clearly displayed along with an image and description of the product. The selection of products will vary based on the particular regulatory scenario that is being modeled. Tobacco and nicotine products will match the products found by surveying product availability vendors in the local communities. In each pricing scenario during each marketplace session, participants will be asked to make nicotine-product purchases sufficient for one week's use from this marketplace. During a purchasing session, the participant will be provided with a virtual budget that matches their actual weekly budget for nicotine/tobacco products, a procedure we have shown to generate realistic results. They will use that virtual budget to indicate which selection of products they would purchase from those available in the marketplace.

Baseline Assessment Session. The first experimental session will be an assessment session to collect information from participants on substance use patterns and addiction severity, as well as the results of behavioral and cognitive tasks that have measure components of our behavioral economic model of product valuation.

Sampling Period. After their assessment session, participants will be given a supply of their randomly assigned reduced-nicotine cigarette corresponding to two weeks of their typical cigarette consumption and asked to use the provided cigarettes as their only combusted tobacco product for 9 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Consume nicotine and/or tobacco products daily
* Have no plans to quit nicotine/tobacco consumption or seek treatment in the subsequent 9 weeks
* Read and understand English

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 473 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Aggregate behavioral economic demand across all participants under the proposed regulatory environments | Assessed at study week 0 and at study week 9
  Participants will complete trials of the Experimental Tobacco Marketplace wherein the price of a target commodity will be increased. Nonlinear mixed effects modeling will be used to fit a curve to estimate the number of products purchased at each price and the analysis will result in an measure of overall price sensitivity under each of the regulatory conditions.
Aggregate behavioral economic substitution across all participants under the proposed regulatory environments | Assessed at study week 0 and at study week 9
  Participants will complete trials of the Experimental Tobacco Marketplace wherein the price of alternative products will be fixed across trials and their usual product will change price. Mixed effects modeling will be used to fit a curve to estimate the slopes and intercepts of these alternative products, revealing the degree to which participants will choose to purchase each alternative product as the price of the participant's usual product increases.

SECONDARY OUTCOMES:
Timeline Follow-Back (TLFB): Average of marijuana and nicotine use quantity | Assessed at study week 0 and at study week 9
  Self-reported marijuana and nicotine product use separated by product type and flavor for the past 60 days.
Fagerström Test for Nicotine Dependence (FTND) | Assessed at study week 0 and at study week 9
  Measure of dependence symptoms, measured on a scale of 0 to 10. A higher score indicates a higher physical dependence on nicotine.
Minnesota Nicotine Withdrawal Scale (MNWS) | Assessed at study week 0 and at study week 9
  Assesses Withdrawal Symptoms. Scored on an ordinal scale ranging from 0 to 3. A higher score indicates increased intensity of symptoms.
Hypothetical quantity purchased in purchase tasks | Assessed at study week 0 and at study week 9
  Measures valuation by assessing hypothetical consumption across a price range and across the range of products used by participants in the past 60 days.
Delay Discounting Tasks | Assessed at study week 0 and at study week 9
  Assesses valuation for future money and nicotine products.
Activity Level Questionnaire - Substance Use Version (ALQ-SUV) | Assessed at study week 0 and at study week 9
  Measures past-month reinforcement from substance-related and substance-free activities, yielding a reinforcement ratio quantifying the proportion of overall reinforcement obtained from nicotine use. The ratio ranges from 0 to 1, with a higher score indicating a greater proportion of reinforcement received from drug-related activities relative to total reinforcement.
Breath Carbon Monoxide (CO) | Collected twice daily through the 10 week duration of the study
  Breath carbon monoxide readings collected using our app
Salivary Cotinine | Collected with assessment sessions at study weeks 0 and 9, as well as twice weekly remotely during interim sampling period
  Salivary cotinine collected with rapid test, verified via smartphone app
Self-reported nicotine product use | Collected daily from study week 1 to study week 9
  The number of tobacco cigarettes, marijuana cigarettes, and other nicotine/tobacco products consumed. Will be collected with our app.
Self-reported withdrawal symptom severity | Collected daily from study week 1 to study week 9
  On a scale from 0 to 9, participants will report their withdrawal symptom severity in our smartphone app. A higher score indicates more severe symptoms.
Self-reported nicotine craving intensity | Collected daily from study week 1 to study week 9
  On a scale from 0 to 9, participants will report their nicotine craving intensity in our smartphone app. A higher score indicates more intense cravings.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified data will be shared.